CLINICAL TRIAL: NCT03547479
Title: Combined Phone Based Video DOT and Mobile Payments for TB Treatment in Cambodia
Brief Title: VDOT and Mobile Payments in Cambodia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI is no longer at the University
Sponsor: University of Southern California (Other)
Collaborators: Operation ASHA (Unknown); National University of Singapore (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Principal Investigator, Michelle Cullen, Research Compliance Manager, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TW010592-01
Record Dates: First submitted 2018-05-22; First posted 2018-06-06 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Intervention Model Description: The study design consists of (a) 4 qualitative focus groups (b) a pretest of 10 patient (c) a pilot randomised study of 60 patients and (d) interviews of stakeholders including healthcare professionals and policymakers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Participants receive current standard of care (DOTS)
- VDOT only (Experimental): Participants receive daily DOTS treatment with video-enabled mobile monitoring, but also maintain regular supervisory checks
  Interventions: Behavioral: VDOT
- VDOT + mobile money incentives (Experimental): Participants receive daily DOTS treatment with video-enabled mobile monitoring supplemented with mobile money incentives, but also maintain regular supervisory checks
  Interventions: Behavioral: VDOT + mobile money

INTERVENTIONS:
Behavioral: VDOT — In VDOT, reminder notifications are sent x minutes prior to the scheduled pill time, and continue every y minutes until the user sends a video of themselves taking their pill via the app. Instructions will be provided in Khmer. The web system has an administrator component whereby a healthcare provider can log in via the Internet to monitor and validate all the videos received that day, and reasons for non-submission.
  Arms: VDOT only
Behavioral: VDOT + mobile money — The VDOT intervention above will be paired with financial incentives in the form of mobile payments in one of the experimental arms.
  Arms: VDOT + mobile money incentives

SUMMARY:
This project proposes to develop and pilot a novel smart phone-based intervention to improve tuberculosis (TB) treatment adherence in Cambodia, which integrates video-enabled Directly Observed Treatment (vDOT) with an automated rewards system that transfers mobile money and eventual phone ownership to compliant patients. The results will be of immediate relevance to Cambodia's National TB Control Program (which is partnering with us), the major implementing field partner Operation ASHA (a leading TB-focused nonprofit organization), as well as other TB control programs seeking new alternatives to improving adherence, especially where traditional DOT may be infeasible or costly, and outside the area of TB where adherence to treatment is critical, such as HIV, and will provide key insights into mobile health (mHealth) programs in a setting relevant to other developing countries. The project will involve building new capacity in Cambodia for behavioral research, mHealth,and communications through hands-on training for study staff in-country, and through general training sessions for internal and external stakeholders.

DETAILED DESCRIPTION:
Tuberculosis (TB) remains one of the leading causes of death from infectious disease worldwide, and treatment adherence a persistent challenge. This is particularly pressing in high-burden, low-resource settings such as Cambodia, where approximately two-thirds of people carry the TB bacterium, one of the highest rates in the world. The investigators propose to develop and pilot a novel smart phone-based intervention to improve TB treatment adherence, integrating video-enabled Directly Observed Therapy (VDOT) with transfers of mobile money and phone ownership to compliant patients. This intervention aims to directly address two of the key barriers to TB treatment adherence in low resource settings where DOT is costly or impractical. First, the video component has the potential to substitute direct in-person observation with time-stamped videos of patients taking their medication. Second, the proposed intervention incorporates incentives to patients for treatment adherence and equipment preservation in the form of mobile money and eventual phone ownership upon treatment completion.

In partnership with the National Tuberculosis Program (NTP), the investigators will assess the feasibility of this intervention and of a future randomized study in two districts of Cambodia. First, the team will extend and adapt an existing platform for video-enabled medication monitoring (Mobile Interactive Supervised Therapy (MIST)) to incorporate mobile cash payments conditional upon compliance. Outstanding technical and usability issues with the platform will be identified and addressed by conducting an initial 1-month test of the intervention with 10 TB patients. Finally, the investigators will conduct an 8-month demonstration study among 50 households in our study locations to assess the acceptability, implementation, and potential for scale up of the intervention. We also aim to assess the practicalities and challenges of a future randomized controlled effectiveness and cost-effectiveness trial.

To the best of our knowledge, this study is the first to examine a mHealth intervention for TB that integrates both adherence monitoring and patient incentives into a single platform. The results will be of immediate relevance to the NTP as well as other TB control programs seeking new alternatives to improving adherence, especially where traditional DOT may be infeasible or costly. These results will also be of interest outside the area of TB where adherence to treatment is critical, such as HIV. More generally, the study will provide key insights into mHealth programs in a setting relevant to other developing countries. This project will involve building new capacity in Cambodia for behavioral research, mHealth, and communications through training to the study personnel and general training on conducting TB and/or mHealth research to study partners and other stakeholders in the country.

ELIGIBILITY:
PROPOSED PATIENT INCLUSION CRITERIA

1. Age 21 years or more;
2. Diagnosis of TB at healthcare facility (Clinical symptoms consistent with pulmonary TB and sputum test positive);
3. Willing to comply with the study procedures;
4. Resident at a fixed address within feasible travelling distance to the site and likely to remain resident there for the foreseeable future;
5. Willing to have directly observed therapy;
6. Willing and able to provide written informed consent in English/Khmer.

PROPOSED PATIENT EXCLUSION CRITERIA

1. Extra-pulmonary TB or suspected rifampicin resistance;
2. Underlying serious chronic diseases (such as liver or kidney disease, active malignancy, poorly-controlled diabetes);
3. History of myocardial infarction, congestive cardiac failure, cardiac arrhythmias or family history of Long QT Syndrome;
4. Current alcohol or drug abuse;
5. Pregnancy;
6. Inability to take oral medication or known allergy to one or more of the study drugs.
7. Any other significant condition that would, in the opinion of the investigator, compromise the patient's safety or outcome in the trial or lead to poor compliance with study visits and protocol requirements;

   -

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2019-05 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility: % patients correctly using the system | 6 months
  % patients correctly using the system without phone theft, breakages or discrepancies in incentive distribution

SECONDARY OUTCOMES:
Missed treatment | 6 months
  Any missed treatment for 10 subsequent days or more
Compliance | 6 months
  Number of pills taken relative to total prescribed
Treatment default | 6 months
  Missed treatment for 2 subsequent months or more
Cure | 5 and 8 months
  Sputum smear-conversion at month 5 and 8

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Yoong, Principal Investigator — University of Southern California

IPD SHARING:
Plan to Share IPD: No